CLINICAL TRIAL: NCT04719494
Title: Dynamic Balance Training in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marquette University (Other)
Collaborators: Greater Milwaukee Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 74915
Record Dates: First submitted 2020-09-04; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training Group (Experimental): During the 12-training day sessions, subjects will walk on the treadmill for a total of 30 minutes. Participants will walk at a comfortable pace while we perform controlled movements to the treadmill system. Subjects will be fitted with a fall-arrest harness and assisted onto the treadmill system. In the dynamic balance training group, we will move the motion base as participants walk in order to challenge their balance.
  Interventions: Other: Dynamic balance walking training
- Control Group (No Intervention): Subjects who are in the control group will also walk on the treadmill, but the motion base will remain stationary. They will complete 12-training day sessions.

INTERVENTIONS:
Other: Dynamic balance walking training — Participants in the training group will walk on an elevated treadmill that will move side-to-side in a pseudorandom manner, thereby increasing the difficulty to their balance. Participants are asked to walk independently for 30-minutes per session, for 12 days over 4 weeks.
  Arms: Training Group

SUMMARY:
This study will test a new technique for improving balance while walking in people with multiple sclerosis (MS). The technique focuses on having people with MS safely practice walking on simulated, uneven terrain that challenges balance and more accurately mimics walking in the community. The goal is to improve balance while walking in order to improve mobility and decrease the risk of falls. Recently, we developed a state-of-the-art treadmill system that allows us to create a challenging walking environment by placing a treadmill onto a motion base. We are able to simulate uneven terrain through movements of the walking surface while maintaining a safe walking environment. We will use this system to conduct tests of balance while walking and to train people to walk on uneven surfaces. Our objective is to evaluate the use of uneven terrain for training gait and balance in people with MS. Participants will undergo a four-week training protocol designed to disrupt and challenge balance while walking. We anticipate that training on uneven terrain will enhance gait stability, improve overall walking function and balance and increase balance confidence compared to training on a stable surface.

ELIGIBILITY:
Inclusion Criteria:

* Participants have been clinically diagnosed with multiple sclerosis
* Must be capable of walking 10 meters independently with no physical assistance
* Must be able to ascend/descend a small staircase (5 steps)
* Medically stable
* Able to give informed consent

Exclusion Criteria:

* they suffer from cognitive deficits that prevent them from following 1 step commands
* unable to give informed consent
* if they suffer from significant cardiovascular problems, respiratory failure, major orthopedic problems, or other medical conditions that affect balance (e.g. diabetic neuropathy, myopathy, or vertigo)
* Significant medical comorbidity or concurrent illness limiting their capacity to conform to study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Change in Functional Gait Assessment | Before and after training (occurs within 5-week period)
  The functional gait assessment (FGA) is a clinically accepted tool and is used to measure postural stability before and after the proposed walking paradigm.
Change in Dynamic Stability | Before and after training (occurs within 5-week period)
  Dynamic Stability is assessed using the margin of stability (MoS). The MoS is defined as the center of mass position and velocity relative to the edge of the person's base of support. If the center of mass falls outside the base of support, the individual may require corrective action to restore balance and/or be at higher risk for loss of balance. For this study, we measured the center of mass motion and foot placement (i.e., base of support) in the medio-lateral direction to calculate each person's MoS before and after the 4-week walking sessions.
Change in Step Width | Before and after training (occurs within 5-week period)
  Step width was measured for all individuals as the distance (centimeters) between the left and right ankle during double-limb support of each gait cycle. We measured step width before and after the 4-week walking sessions.

SECONDARY OUTCOMES:
Change in Step Length | Before and after training (occurs within 5-week period)
  Step Length was measured for all individuals as the distance (centimeters) between the left big toe and right big toe at the time the heel of the leading foot made contact with the treadmill belt at each gait cycle. We measured step length before and after the 4-week walking sessions.
Change in Step Frequency | Before and after training (occurs within 5-week period)
  Step Frequency was measured for all individuals as the number of steps occurring within a 60-second time window (units of Hz). We measured step frequency before and after the 4-week walking sessions.
Change in 10-Meter Walk Test | Before and after training (occurs within 5-week period)
  The 10-Meter Walk Test was administered at self-selected overground walking speeds for each individual. We assess walking speed with this tool before and after the proposed walking paradigm.

IPD SHARING:
Plan to Share IPD: No